CLINICAL TRIAL: NCT04525898
Title: Intraoperative Methadone for Postoperative Pain Control After Thoracic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EH19-031
Record Dates: First submitted 2020-02-12; First posted 2020-08-25 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone

STUDY DESIGN:
Intervention Model Description: One group of patients will be randomized to receive a dose of methadone at induction of anesthesia (0.15 mg/kg ideal body weight (IBW)-methadone group)). The other group will be randomized to be administered an equal volume of saline in an identical appearing syringe (control group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The hospital pharmacy will prepare two identical-appearing syringes; one will contain methadone and the other saline. The patients, care providers, and researchers will all be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone Group (Active Comparator): The methadone group will receive a dose of methadone at induction of anesthesia (0.15 mg/kg ideal body weight (IBW)
  Interventions: Drug: Methadone
- Control Group (Placebo Comparator): The control group will be administered an equal volume of saline in an identical appearing syringe.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — The methadone group will receive an intravenous dose of methadone at induction of anesthesia (0.15 mg/kg ideal body weight (IBW)

SUMMARY:
Pain following surgery continues to be an important adverse outcome that may impact postoperative recovery. Opioids like fentanyl and hydromorphone are the primary medications used to provide analgesia, but paradoxically, may actually worsen pain when administered in the operating room. Methadone is a unique opioid which has N-methyl-D-aspartate (NMDA) receptor blocking properties, which may prevent the development of opioid-induced tolerance and hyperalgesia (increased sensitivity to pain induced by a drug). Studies have demonstrated that methadone reduces the need for analgesic medications and decreases pain after surgery. Furthermore, the addition of methadone to a standard anesthetic has been demonstrated to increase patient satisfaction with pain management and reduce the need for opioid analgesic medications during the first month after surgery. Some investigators have described methadone as a "opioid-sparing opioid" and recommended its use as part of a multimodal pain management strategy.

There is a growing interest in reducing the use of traditional opioids in the operating room. The aim of this clinical trial is to compare pain scores and analgesic requirements in two groups of patients; one group will be randomized to receive a small dose of methadone at the start of surgery. The other group will be randomized to receive an equal volume of saline (salt water-control group) at the start of surgery. We hypothesize that patients randomized to be administered methadone at the start of surgery will have less postoperative pain and may require lower doses of pain medications than those given saline-control..

DETAILED DESCRIPTION:
Despite the development of a number of treatment strategies for pain after surgery, many patients continue to experience moderate-to-severe pain in the early postoperative period. Traditionally, opioids are the primary method of providing analgesia in the operating room, postanesthesia care unit (PACU), intensive care unit, and surgical wards. However, a number of potentially life-threatening complications can develop following opioid administration including severe respiratory depression. In addition, studies have demonstrated an association between the dose of opioid used in the operating room and the intensity of pain after following surgery; paradoxically, the greater the dose of opioid administered, the higher the reported pain scores are in the early recovery period. This is likely secondary to two interrelated phenomena: tolerance and opioid-induced hyperalgesia. Tolerance, a pharmacologic concept, can develop acutely after a single dose of opioid in the operating room. This can result in increased requirements for postoperative pain medications. Opioid-induced hyperalgesia (OIH), a clinical concept, involves enhancement of existent pain stimuli (normally minimally painful incisions may feel much worse) and facilitation of chronic pain development. Therefore, it may be beneficial to use lower doses of intraoperative opioids on all surgical patients.

Using a multimodal approach to pain management has been demonstrated to reduce the requirements for postoperative analgesic agents and improve pain scores. A number of different agents have been investigated including gabapentinoids, lidocaine, steroids, and nonsteroidal anti-inflammatory agents. Although it is an opioid, another medication that may be considered as part of a multimodal treatment of pain is methadone. Methadone has several unique properties that may beneficially impact the recovery of the surgical patient. It has been extensively studied as an agent to provide prolonged postoperative analgesia. When larger doses of methadone have been administered intravenously at induction of anesthesia, a median duration of analgesia lasting more than 25 hours has been reported. In patients undergoing abdominal, orthopedic, or gynecologic surgery, the use of a single dose of methadone (20 mg or 0.2-0.3 mg/kg) before surgical incision resulted in improved analgesia for the first 24-48 hours after surgery, when compared to other intraoperative opioids. In these investigations, patients in the methadone groups required significantly less postoperative pain medication and reported lower pain scores during the first or second postoperative days. However, other investigations have demonstrated significant analgesic effects of smaller doses of methadone (0.1 to 0.15 mg/kg). Furthermore, reductions in pain scores and need for oral opioid medications for the first 30 postoperative days have been observed in surgical patients administered 0.15 mg/kg of methadone. In addition to a long plasma half-life, methadone has other properties which may be advantageous in surgical patients. Recent evidence has demonstrated that methadone has the ability to block N-methyl-D-aspartate (NMDA) receptors. NMDA receptors have been implicated in the development of postoperative hyperalgesia (amplification of pain stimuli), and techniques which block NMBA receptors reduce pain. Therefore, methadone may attenuate postoperative pain via this additional mechanism. NMDA receptor stimulation is also thought to play an important role in the development of chronic pain. Although unproven, it has been hypothesized that methadone may reduce the risk of development of chronic postsurgical pain via inhibition of NMDA receptors. No adverse events directly attributable to methadone have been reported in any of the published clinical trials.

The aim of this randomized clinical investigation is to assess two cohorts of patients; one group will receive a dose of methadone at induction of anesthesia (0.15 mg/kg ideal body weight (IBW)-methadone group)). The other group will be randomized to be administered an equal volume of saline in an identical appearing syringe (control group).. The primary endpoint will be pain scores 24 hours after surgery. Secondary endpoints will include pain scores on arrival and discharge from the postanesthesia care unit (PACU), and at 2, 6, 24, 48, and 72 hours (if the patient remains in the hospital) after surgery. Analgesic requirements in the PACU and surgical wards will be assessed. In addition, the incidence of potential methadone-related side effects will be measured (delayed emergence, nausea and vomiting, respiratory depression)). Furthermore, methadone has been documented to potentially reduce the incidence of chronic postsurgical pain. A survey with a self-addressed stamped envelope will be provided to patients at 1, 3, 6, and 12 months after surgery to complete to assess the effect of methadone on this important outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing any thoracoscopic procedure under general anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists Physical Status 4 or 5, active heart failure, significant liver disease, previous adverse reactions to methadone, preoperative recent history of opioid or alcohol abuse, renal failure, or inability to comprehend the English language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 24 hours after thoracic surgery
  Pain scores 24 hours after the surgical procedure

SECONDARY OUTCOMES:
Pain Scores | 2 hours after thoracic surgery
  Pain scores 2 hours after the surgical procedure
Pain Scores | 6 hours after thoracic surgery
  Pain scores 6 hours after the surgical procedure
Pain Scores | 48 hours after thoracic surgery
  Pain scores 48 hours after the surgical procedure
Pain Scores | 72 hours after thoracic surgery
  Pain scores 72 hours after the surgical procedure
Analgesic requirements | At 24 hours
  Postoperative opioid needs
Analgesic requirements | At 48 hours
  Postoperative opioid needs
Chronic Pain | 1 month
  Pain intensity after surgical discharge-Pain assessed at rest and with coughing on a 0 to 10 scale with 0=no pain and 10=worst pain imaginable
Chronic Pain | 3 months
  Pain intensity after surgical discharge-Pain assessed at rest and with coughing on a 0 to 10 scale with 0=no pain and 10=worst pain imaginable
Chronic Pain | 6 months
  Pain intensity after surgical discharge--Pain assessed at rest and with coughing on a 0 to 10 scale with 0=no pain and 10=worst pain imaginable
Chronic Pain | 12 months
  Pain intensity after surgical discharge--Pain assessed at rest and with coughing on a 0 to 10 scale with 0=no pain and 10=worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data not to be shared